CLINICAL TRIAL: NCT05180630
Title: Sound Quality and Occlusion Comparisons With Different Hearing Aid Couplings and Venting Systems
Brief Title: Sound Quality Comparisons With Different Hearing Aid Couplings and Venting Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SRF-465
Record Dates: First submitted 2021-11-25; First posted 2022-01-06 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Custom earmolds, then Open domes, then Vented domes (Experimental): Participants first fit with Audeo 90P hearing aids and custom earmolds with dynamic venting, then fit with the same hearing aids using open domes, then fit with the same hearing aids using vented domes.
  Interventions: Device: Audeo P90 hearing aid with custom earmolds using dynamic venting; Device: Audeo P90 hearing aid with Open domes; Device: Audeo P90 hearing aid with Vented domes
- Open domes, then Vented domes, then Custom earmolds (Experimental): Participants first fit with Audeo 90P hearing aids and open domes, then fit with the same hearing aids using vented domes, then fit with the same hearing aids using custom earmolds with dynamic venting.
  Interventions: Device: Audeo P90 hearing aid with custom earmolds using dynamic venting; Device: Audeo P90 hearing aid with Open domes; Device: Audeo P90 hearing aid with Vented domes
- Vented domes, then Custom earmolds, then Open domes (Experimental): Participants first fit with Audeo 90P hearing aids and vented domes, then fit with the same hearing aids using custom earmolds with dynamic venting, then fit with the same hearing aids using open domes.
  Interventions: Device: Audeo P90 hearing aid with custom earmolds using dynamic venting; Device: Audeo P90 hearing aid with Open domes; Device: Audeo P90 hearing aid with Vented domes

INTERVENTIONS:
Device: Audeo P90 hearing aid with custom earmolds using dynamic venting — Audeo P90 hearing aids coupled to custom earmolds that use dynamic venting.
Device: Audeo P90 hearing aid with Open domes — Audeo P90 hearing aid coupled with non-custom, manufacturer open domes
Device: Audeo P90 hearing aid with Vented domes — Audeo P90 hearing aid coupled with non-custom, manufacturer vented domes

SUMMARY:
Participants will be comparing the sound quality of their own voice and the sound quality of streamed music using universal couplings and a custom earmold with a dynamic vent.

ELIGIBILITY:
Inclusion Criteria:

* Mild to severe bilateral sensorineural hearing loss
* hearing must be symmetrical below 500 Hz
* must live within 30 miles of Aurora IL

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova US, Aurora, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Custom Earmolds, Then Open Domes, Then Vented Domes: Participants first fit with Audeo 90P hearing aids and custom earmold with dynamic venting, then fit with the same hearing aids using open domes, then fit with the same hearing aids using vented domes.
Period: First Intervention
Arm/Group | Custom Earmolds, Then Open Domes, Then Vented Domes | Open Domes, Then Vented Domes, Then Custom Earmolds | Vented Domes, Then Custom Earmolds, Then Open Domes
Started | 6 | 6 | 5
Completed | 6 | 6 | 2
Not Completed | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 3
Period: Second Intervention
Arm/Group | Custom Earmolds, Then Open Domes, Then Vented Domes | Open Domes, Then Vented Domes, Then Custom Earmolds | Vented Domes, Then Custom Earmolds, Then Open Domes
Started | 6 | 6 | 2
Completed | 6 | 6 | 2
Not Completed | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Custom Earmolds, Then Open Domes, Then Vented Domes | Open Domes, Then Vented Domes, Then Custom Earmolds | Vented Domes, Then Custom Earmolds, Then Open Domes
Started | 6 | 6 | 2
Completed | 6 | 6 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Group: Group will be fit using three different hearing aid couplings. Each participant will be supplying a rating of sound quality for each condition.
  Audeo P90 hearing aid with compatible couplings: Audeo P90 hearing aids will be fit with three different compatible couplings.
Arm/Group | Study Group
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: years] | 71 [59 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14
Mild to moderate hearing loss [Count of Participants; unit: Participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: Sound Quality of Streamed Music Rating Scale
Description: subjective rating on scale from 0 (worst) to 100 (best) for sound quality of streamed signal
Time Frame: 1 day
Population: All participants who evaluated the sound quality of streamed music using all three coupling systems.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Custom Earmolds, Then Open Domes, Then Vented Domes | Open Domes, Then Vented Domes, Then Custom Earmolds | Vented Domes, Then Custom Earmolds, Then Open Domes
Number analyzed (Participants) | 6 | 6 | 2
score on a scale
  Subjective sound quality rating of streamed music with custom earmolds | 84 [75 to 100] | 70 [25 to 100] | 70 [60 to 80]
  Subjective sound quality rating of streamed music using open domes | 90 [80 to 100] | 62.5 [25 to 100] | 80 [70 to 90]
  Subjective sound quality rating of streamed music using vented domes | 94 [84 to 100] | 81 [50 to 100] | 90 [80 to 100]
Statistical Analysis 1: Comparison: Custom Earmolds, Then Open Domes, Then Vented Domes vs Open Domes, Then Vented Domes, Then Custom Earmolds vs Vented Domes, Then Custom Earmolds, Then Open Domes; Treatment order was not analyzed. A repeated measures ANOVA was performed to compare the effect of the coupling conditions on sound quality ratings for streamed music, but there was no analysis between groups; Test type: Other; p = 0.012, ANOVA — When p-value is adjusted for multiple comparisons, the level of statistical significance must be </= to 0.01666667 (.05/3). Comparisons were total mean scores for Open dome condition, Vented dome condition, and Custom earmolds with dynamic venting

2. Primary Outcome: Own Voice Sound Quality Rating Scale
Description: subjective rating on a scale from 0 (worst) to 100 (best) for sound quality of participant's own voice quality.
Time Frame: 1 day
Population: All participants who rated sound quality of own voice using hearing aids with all three coupling systems.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Open Domes, Then Vented Domes, Then Custom Earmolds: Participants first fit with Audeo 90P hearing aids and open domes then fit with the same hearing aids using vented domes, then fit with the same hearing aids using custom earmolds with dynamic venting.
Arm/Group | Custom Earmolds, Then Open Domes, Then Vented Domes | Open Domes, Then Vented Domes, Then Custom Earmolds | Vented Domes, Then Custom Earmolds, Then Open Domes
Number analyzed (Participants) | 6 | 6 | 2
score on a scale
  Subjective rating of own voice using custom earmolds with dynamic venting | 69.2 [50 to 90] | 75 [55 to 90] | 40 [30 to 50]
  Subjective rating of own voice sound quality using open domes | 80 [63 to 98] | 78 [50 to 100] | 50 [25 to 75]
  Subjective rating of own voice sound quality using vented domes | 85 [75 to 100] | 73 [40 to 100] | 65 [55 to 75]
Statistical Analysis 1: Comparison: Custom Earmolds, Then Open Domes, Then Vented Domes vs Open Domes, Then Vented Domes, Then Custom Earmolds vs Vented Domes, Then Custom Earmolds, Then Open Domes; Treatment order was not analyzed. A repeated measures ANOVA was performed to compare the effect of the coupling conditions on sound quality ratings for own voice, but there was no analysis between groups; Test type: Other; p = 0.154, ANOVA — When p-value is adjusted for multiple comparisons, the level of statistical significance must be </= to 0.01666667 (.05/3)

ADVERSE EVENTS:
Time Frame: Two separate appointments, one day each, for a total of two non-consecutive days.
Groups:
- Participants Who Received Intervention of Custom Earmolds With Dynamic Venting: All participants who received the intervention of custom earmolds with dynamic venting.
- Participants Who Received Intervention of Open Domes: All participants who received the intervention of open domes.
- Participants Who Received Intervention Vented Domes: All participants who received the intervention of vented domes.
Arm/Group | Participants Who Received Intervention of Custom Earmolds With Dynamic Venting | Participants Who Received Intervention of Open Domes | Participants Who Received Intervention Vented Domes
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT05180630/Prot_SAP_001.pdf